CLINICAL TRIAL: NCT02979028
Title: The Protective Effect of Transcutaneous Electrical Acupoint Stimulation (TEAS) on Aged Patients Undergoing Lower Extremity Arthroplasty: A Single-Center, Double-Blinded, Randomised Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation (TEAS) on Aged Patients Undergoing Lower Extremity Arthroplasty
Acronym: TEAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: zxy
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2016-11

CONDITIONS: Joint Replacement
Keywords: TEAS; complication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TEAS group (Experimental): Electric stimulation was given through electrode attached to acupoints SP6 and ST36 .TEAS will be administered 30 minutes prior to surgery and continued until the end of the surgery.
  Interventions: Device: TEAS
- Sham group (Sham Comparator): Non-acupoint is located 2cm inward to the specific acupoints.TEAS will be administered 30 minutes prior to surgery and continued until the end of the surgery.
  Interventions: Device: TEAS
- Control group (Placebo Comparator): Control patients will receive the same treatment without electrical stimulation.
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS — Transcutaneous electrical acupoint stimulation

SUMMARY:
This is a single center, randomized, double-blinded, controlled clinical trial. The purpose of this study is to to determine whether treating by transcutaneous electrical acupoint stimulation (TEAS) during perioperative could alleviate the postoperative complications in patients undergoing artificial joint replacement surgery.

DETAILED DESCRIPTION:
The complications from patients accepted artificial joint replacement surgery will directly or indirectly affect the prognosis of the patients, resulting in patients with delayed recovery and increase the hospitalization time and cost. Serious complications can lead to patients deaths during perioperative period. It has been proved that the electroacupuncture application during perioperative period can reduce the dosage of anesthetic drugs, and has a good effect on the protection of the heart and brain. At the same time, the electroacupuncture can also regulate the body's immune function, reduce allergy, reduce postoperative pain and so on.Compared with acupuncture, transcutaneous electric acupoint stimulation (TEAS) is a noninvasive technique that has similar effects to acupuncture. The investigators hypothesize that TEAS before anesthesia and during surgery would decrease the morbidity and mortality of postoperative complications in 30 days after artificial joint replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ASAⅡ-Ⅲ,elective operation patients
2. No other severe complications history
3. Able to give informed consent

Exclusion Criteria:

1. Having severe comorbidity resulting in estimated life expectancy <1 year.
2. Infection at the electroacupuncture site.
3. Suffered from neurologic disorder or impaired mental state
4. Participate in the other clinical trial 3 months before the enrollment
5. No suitable to participate in this experiment

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative complications | within 30 days after operation
  Participants will be followed for the incidence of postoperative complications

SECONDARY OUTCOMES:
length of postoperative hospital stay | an expected average of 1 week
  Participants will be followed for the duration of hospital stay
Quality of life during 30 days after surgery | One month
  evaluate the quality of life after surgery by WHO QOL-BREF scale with interview ，WHO QOL-BREF scale includes five aspects: physical, psychological, social, environmental, integrated, divided into five levels
ICU transfer rate after operation | One month
  Participants will be followed for ICU transfer rate after operation

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Guo, Study Chair — Second Hospital of Shanxi Medical University

REFERENCES:
- [Background] Huddleston JI, Maloney WJ, Wang Y, Verzier N, Hunt DR, Herndon JH. Adverse events after total knee arthroplasty: a national Medicare study. J Arthroplasty. 2009 Sep;24(6 Suppl):95-100. doi: 10.1016/j.arth.2009.05.001. Epub 2009 Jul 4. PMID 19577884
- [Background] Geerts WH, Pineo GF, Heit JA, Bergqvist D, Lassen MR, Colwell CW, Ray JG. Prevention of venous thromboembolism: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):338S-400S. doi: 10.1378/chest.126.3_suppl.338S. PMID 15383478
- [Background] Singh JA, Jensen MR, Harmsen WS, Gabriel SE, Lewallen DG. Cardiac and thromboembolic complications and mortality in patients undergoing total hip and total knee arthroplasty. Ann Rheum Dis. 2011 Dec;70(12):2082-8. doi: 10.1136/ard.2010.148726. Epub 2011 Oct 21. PMID 22021865
- [Background] Krecisz B, Kiec-Swierczynska M, Chomiczewska-Skora D. Allergy to orthopedic metal implants - a prospective study. Int J Occup Med Environ Health. 2012 Sep;25(4):463-9. doi: 10.2478/S13382-012-0029-3. Epub 2012 Dec 3. PMID 23212287
- [Background] Hou L, Chen C, Xu L, Yin P, Peng W. Electrical stimulation of acupoint combinations against deep venous thrombosis in elderly bedridden patients after major surgery. J Tradit Chin Med. 2013 Apr;33(2):187-93. doi: 10.1016/s0254-6272(13)60123-5. PMID 23789215
- [Background] Yang L, Yang J, Wang Q, Chen M, Lu Z, Chen S, Xiong L. Cardioprotective effects of electroacupuncture pretreatment on patients undergoing heart valve replacement surgery: a randomized controlled trial. Ann Thorac Surg. 2010 Mar;89(3):781-6. doi: 10.1016/j.athoracsur.2009.12.003. PMID 20172127
- [Background] Ni X, Xie Y, Wang Q, Zhong H, Chen M, Wang F, Xiong L. Cardioprotective effect of transcutaneous electric acupoint stimulation in the pediatric cardiac patients: a randomized controlled clinical trial. Paediatr Anaesth. 2012 Aug;22(8):805-11. doi: 10.1111/j.1460-9592.2012.03822.x. Epub 2012 Mar 2. PMID 22380768